CLINICAL TRIAL: NCT00352729
Title: Evaluation of ACell Hydrated Wound Dressing for Autogenous Skin Donor Sites
Acronym: ACell
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI decided to use another product
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Leopoldo Cancio, LTC, MC, USAISR
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-06-002
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Burns
Keywords: Burns; ACell; Donor Site
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator)
  Interventions: Device: ACell dressing

INTERVENTIONS:
Device: ACell dressing — dressing

SUMMARY:
The purpose of this study is to see if treating a donor site wound with the ACell dressing is as good as or better than the dressings we currently treat harvested donor sites with. This will be tested on consenting burn patients who require excision and grafting surgery for their burn wounds.

Hypothesis: The mean healing time for wounds treated with the ACell dressing will be less than the mean healing time for wounds treated with the Standard of Care dressing.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, and controlled study to evaluate the effectiveness of the ACell Dressing for use as a dressing for autogenous skin donor sites compared to our current standard donor site dressing, which is currently Xeroform.

ELIGIBILITY:
Inclusion Criteria:

* less than 30% total body surface area burn
* burn wounds do not involve the donor site harvesting areas
* requires excision and grafting of sufficient extent to justify two donor site of roughly equal size on non-dependent body surfaces.
* The scheduled excision and grafting procedure is the first such operation for the subject
* subject agrees to participate in follow-up evaluations

Exclusion Criteria:

* Critical illnesses such as those requiring ventilator support, systemic infection, or hemodynamic instability
* Major acute or chronic medical illness that could affect wound healing
* Cellulitis or other infection of the potential donor sites
* Donor site has been previously harvested for grafting
* Subjects who are pregnant
* Religious objections or allergy to porcine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The specific aim of this study is to determine if the ACell dressing is superior to the ISR Burn Center's current standard of care dressing with respect to speed of healing, patient comfort or wound cosmesis. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Albrecht, MD, Principal Investigator — U.S. Army Institute of Surgical Research
Locations (1):
- U.S. Army Insitute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Badylak SF. Xenogeneic extracellular matrix as a scaffold for tissue reconstruction. Transpl Immunol. 2004 Apr;12(3-4):367-77. doi: 10.1016/j.trim.2003.12.016. PMID 15157928